CLINICAL TRIAL: NCT02379299
Title: Dual-Hormone Closed-Loop Glucose Control in Type 1 Diabetes
Brief Title: DiaCon Dual-Hormone Closed-Loop Glucose Control
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Technical University of Denmark (Other)
Responsible Party: Principal Investigator, Signe Schmidt, MD, Hvidovre University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: DHCL2014
Record Dates: First submitted 2015-02-27; First posted 2015-03-04 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2016-08

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single-hormone closed-loop control (Active Comparator): Closed-loop glucose control by use of insulin only by use of DiaCon single-hormone closed-loop glucose control algorithm
  Interventions: Device: DiaCon single-hormone closed-loop glucose control algorithm
- Dual-hormone closed-loop control (Experimental): Closed-loop glucose control by use of insulin and glucagon by use of DiaCon dual-hormone closed-loop glucose control algorithm
  Interventions: Device: DiaCon dual-hormone closed-loop glucose control algorithm

INTERVENTIONS:
Device: DiaCon dual-hormone closed-loop glucose control algorithm — Dual-hormone closed-loop glucose control
  Arms: Dual-hormone closed-loop control
Device: DiaCon single-hormone closed-loop glucose control algorithm — Single-hormone closed-loop glucose control
  Arms: Single-hormone closed-loop control

SUMMARY:
The ultimate T1D treatment tool is a closed-loop glucose control system, i.e. a fully automated system for intensive insulin treatment. Such system will ease the burden of constant treatment decision-making and at the same time it has the potential to safely intensify insulin therapy such that more patients can reach treatment goals. Currently, no off-the-shelf closed-loop system exists but research efforts in this field have been intensified and resulted in great progress in recent years. Most closed-loop systems consist of an insulin pump, a CGM, and a control algorithm residing on a mobile computer that continuously (every 5-15 min) computes the optimal insulin dosage from the CGM values. For daytime blood glucose control, however, we believe that the system needs to be further advanced. Consequently, we have extended our single-hormone closed-loop system such that it now includes a second pump for glucagon delivery and correspondingly we have further developed our control algorithm to compute both insulin and glucagon dosages.

We hypothesize that we have developed a safe and effective dual-hormone closed-loop system for patients with type 1 diabetes and that this system is superior to single-hormone closed-loop therapy. The aims of this two-phase project are to 1) demonstrate proof-of-concept and 2) to compare dual-hormone with single-hormone closed-loop glucose control.

ELIGIBILITY:
Inclusion Criteria:

* T1D ≥ 2 years
* Insulin pump therapy with rapid-acting analog insulin ≥ 1 year
* HbA1c ≤ 8.5% (69 mmol/mol)
* Ability and willingness to comply with all protocol procedures

Exclusion Criteria:

* Pregnancy or nursing
* Plan to become pregnant or sexually active and not using adequate contraceptive methods (sterilization, intrauterine device, contraceptive pill, patch or injection)
* Hypoglycemia unawareness (self-reported lack of hypoglycemia symptoms when blood glucose is < 3.0 mmol/l)
* Use of anti-diabetic medicine (other than insulin), corticosteroids or other drugs affecting glucose metabolism during or within 30 days prior to study participation
* History of coronary artery disease or congestive heart failure
* Abnormal ECG suggestive of coronary artery disease and increased risk of malignant arrhythmia
* Allergy to glucagon or lactose
* Pheochromocytoma
* Other concomitant medical or psychological condition that according to the investigator's assessment makes the patient unsuitable for study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2017-07-22 (Actual)

PRIMARY OUTCOMES:
Percentage of time with glucose values < 3.9 mmol/l as measured by Continuous Glucose Monitoring and Yellow Spring Instruments | Every 5 minutes for 33 hours (total duration of each study arm)
Number of CHO interventions to treat hypoglycemia | 33 hours (total duration of each study arm)

CONTACTS AND LOCATIONS:
Overall Officials: Signe Schmidt, MD, PhD, Principal Investigator — Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark